CLINICAL TRIAL: NCT05045092
Title: A Follow-up Study of Neonates Receiving Extracorporeal Life Support in China
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Chinese Neonatal Network (Other)
Responsible Party: Sponsor
Other Study IDs: F-NELS
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Extracorporeal Life Support; Neurodevelopment; Neonate; Mortality; Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Descriptive study of two-year follow-up outcomes of surviving neonates who are enrolled in the Chinese Neonatal Extracorporeal Life Support Registry (Chi-NELS) from 2022 to 2024.

DETAILED DESCRIPTION:
This study aims to describe the six -month, one-year and two-year neurodevelopmental outcomes of survivors of neonatal ECLS treatment in the Chi-NELS. The study population will be neonates who receive ECLS support within 28 days of life and are enrolled in the Chi-NELS. These infants will be prospectively followed for two years. Mortality, growth, and neurodevelopmental outcomes will be assessed at six months, one year and two years.

ELIGIBILITY:
Inclusion Criteria:

* Infants who receive extracorporeal life support (ECLS) at ≤28 days of life from 2022.1.1-2023.12.31
* Survive to the first ICU discharge

Exclusion Criteria:

* Infants who died during the ECLS hospitalization
* Parental refusal to follow-up

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates who receive ECLS support within 28 days of life and survive to the first discharge.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality or severe/moderate neurodevelopmental delay at two-year old | At two-year old
  It is a binary variable (1/0). If mortality or severe/moderate neurodevelopmental delay occur in the participent, the value of this varible is 1.

SECONDARY OUTCOMES:
Body weight of infants at six months | At six months
Length of infants at six months | At six months
Head circumference of infants at six months | At six months
Body weight of infants at one year old | At one year old
Length of infants at one year old | At one year old
Head circumference of infants at one year old | At one year old
Body weight of infants at two years old | At two years old
Length of infants at two years old | At two years old
Head circumference of infants at two years old | At two years old
Severe/moderate neurodevelopmental delay at six months | At six months
  Proportion of infants with severe/moderate neurodevelopmental delay according to the development scale
Severe/moderate neurodevelopmental delay at one year old | At one year old
  Proportion of infants with severe/moderate neurodevelopmental delay according to the development scale
Severe/moderate neurodevelopmental delay at two years old | At two years old
  Proportion of infants with severe/moderate neurodevelopmental delay according to the development scale

CONTACTS AND LOCATIONS:
Overall Officials: Yun Cao, Ph.D, M.D., Principal Investigator — Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No